CLINICAL TRIAL: NCT04118946
Title: Intra Vesical Instillation Versus Submucosal Injection of Platelet Enriched Plasma for Treatment of Interstitial Cystitis/Bladder Pain Syndrome: A Randomized Controlled Trial
Brief Title: Platelet Enriched Plasma for Treatment of Interstitial Cystitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Sobhy Elhefnawy, principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.19.03.540
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome; Platelet Enriched Plasma
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Patients with diagnosis of Interstitial cystitis/ Bladder pain syndrome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravesical instillation (Active Comparator): Intravesical instillation of platelet enriched plasma every week for 6 weeks
  Interventions: Biological: platelet enriched plasma
- submucosal injection (Active Comparator): submucosal injectionof platelet enriched plasma
  Interventions: Biological: platelet enriched plasma

INTERVENTIONS:
Biological: platelet enriched plasma — PRP is prepared via a two-step centrifugation preparation of a blood sample, which is cured with an anticoagulant. Then either with be applied through urethral catheter in one arm or via submucos injection in anther one.

SUMMARY:
A prospective randomized trial will be conducted aiming at evaluation the efficacy and safety of platelet enriched plasma for management of bladder pain syndrome .

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of interstitial cystitis/ Bladder painful Syndrome for more than 3 months will be enrolled

Exclusion Criteria:

* Patients with Anemia, blood disorders, history of pelvic irradiation, pelvic malignancy, and active urinary tract infection unless treated, vesical stone, gynecological disorders e.g. uterine fibroid and neurological disorders will be excluded. Patients less than 18 years old will not be allowed to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
efficacy as measured by global response assessment "GRA" | 3 month for each case. Expected time about 18-24 months for whole study period
  It will be measured by global response assessment as main tool. Other measurable outcomes including visual analogue scale for pain, Interstitial Cystitis Symptom Index (4 questions) and Problem Index (4 questions) (ICSI/ICPI). These measures will be collected after each session during period of administration of treatment then at 3 months after end of treatment

SECONDARY OUTCOMES:
safety : rate of complication and grade of complications graded by Dindo-Clavien classification | 3 month for each case. Expected time about 18-24 months for whole study period
  patients will be asked and observed for any anticipated adverse events as hematuria, dysurea, any drug reaction. They will be kept for observation in hospital for 4 hours after delivery for treatment. Periodic reporting of any adverse event by phone call or during next visit.
incidence of urinary tract infection and gynecological infection among this group | 3 month for each case. Expected time about 18-24 months for whole study period
  by doing urine analysis+/- culture if indicated. By doing vaginal swap for culture if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Hefnawy, Msc, MD, Principal Investigator — Assistant professor of urology .Mansoura Urology and Nephrology Center
Locations (1):
- Ahmed S EL Hefnawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No